CLINICAL TRIAL: NCT06926660
Title: A Phase II Randomised, Double-blind, Parallel-group, Multicentre, International Trial to Investigate the Safety and Efficacy of Vicadrostat and Empagliflozin Administered With Simultaneous vs Staggered Initiation in Participants With Chronic Kidney Disease at Risk of Kidney Disease Progression
Brief Title: A Study to Test Whether Vicadrostat in Combination With Empagliflozin Helps People With Chronic Kidney Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1378-0023; 2024-518457-42-00 (Registry Identifier: CTIS); U1111-1314-0083 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-04-11; First posted 2025-04-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo followed by vicadrostat/empagliflozin (Placebo Comparator)
  Interventions: Drug: Vicadrostat; Drug: Empagliflozin; Drug: Placebo matching vicadrostat
- Vicadrostat/empagliflozin (Experimental)
  Interventions: Drug: Vicadrostat; Drug: Empagliflozin

INTERVENTIONS:
Drug: Vicadrostat — Vicadrostat
Drug: Empagliflozin — Empagliflozin
Drug: Placebo matching vicadrostat — Placebo matching vicadrostat
  Arms: Placebo followed by vicadrostat/empagliflozin

SUMMARY:
This study is open to adults with chronic kidney disease (CKD) that is at risk of getting worse. People who have taken a specific type of medication for kidney disease called SGLT2 inhibitor within 1 month before the study or have certain health conditions cannot take part in this study. The purpose of this study is to find out whether a medicine called vicadrostat, used in combination with another medicine called empagliflozin, works in people with chronic kidney disease.

In this study, participants are randomly assigned to one of two groups. Participants have an equal chance of being assigned to either group. In one group, participants take the 2 study medicines, vicadrostat and empagliflozin, every day for 3 months. In the other group, participants take placebo and empagliflozin for the first 1.5 months, and then they take vicadrostat and empagliflozin together for the next 1.5 months. The study medicines are taken orally as tablets. Placebo tablets look like vicadrostat tablets but do not contain any medicine.

Participants are in the study for about 4.5 months. During this time, they visit the study site multiple times. Doctors regularly test kidney function by measuring specific proteins in the blood and urine.

The results are compared between the two groups to see whether there are differences between starting the study medicines at the same time or one after the other. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old and at least of the legal age of consent in countries where it is greater than 18 years.
2. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
3. Male or female participants. Woman of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per International Council on Harmonisation (ICH) M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. For men, birth control is not required during the trial. A list of contraception methods meeting these criteria and instructions on the duration of use is provided in the participant information.
4. Evidence of Chronic Kidney Disease (CKD) at risk of progression based on two Estimated Glomerular Filtration Rate (eGFR) measurements recorded recently (i.e. within 1 year) and at the time of Visit 1, with each Estimated Glomerular Filtration Rate (eGFR) ≥20 and <60 mL/min/1.73m2, irrespective of urine albumin creatinine ratio (UACR). The first of these measurements will be In Approval assessed from historical local laboratory results, and the second will be determined from serum creatinine analysed by the central laboratory at Visit 1.
5. Treatment with a clinically appropriate, stable dose of either Angiotensin-converting enzyme inhibitor (ACEi) or Angiotensin II Receptor Blockers (ARB) (but not both together) for ≥4 weeks before Visit 1, with no planned changes of the therapy for the duration of the trial.

Exclusion Criteria:

1. Treatment with an SGLT2i within 4 weeks before Visit 2. Treatment with a sodium glucose co transporter 2 inhibitor (SGLT2i) should not be interrupted with the intention of enrolment into the trial.
2. Treatment with an mineralocorticoid receptor antagonist (MRA), aldosterone synthase inhibitor (ASi), or potassium-sparing diuretic(s) within 14 days prior to Visit 1, or requiring such treatment before randomisation, or planned during the trial, based on the judgment of the investigator. Treatment with an MRA or ASi should not be interrupted with the intention of enrolment into the trial.
3. Blood potassium of >5.2 mmol/L at Visit 1.
4. Blood Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) >3x Upper limit of normal (ULN) at Visit 1.
5. Known severe hepatic impairment (i.e. Child Pugh class C cirrhosis).
6. On dialysis, functioning kidney transplant, or scheduled for transplant.
7. Treated with new immunosuppression therapy for new (or relapse/flare of pre-existing) kidney disease within the last 60 days.
8. Currently treated with systemic mineralocorticoid replacement therapy (e.g. fludrocortisone).

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2027-01-08 (Estimated); Study Completion 2027-01-08 (Estimated)

PRIMARY OUTCOMES:
Absolute change in estimated glomerular filtration rate (eGFR) (mL/min/1.73m2) from baseline to Week 14 | At baseline, up to week 14

SECONDARY OUTCOMES:
Absolute change in estimated glomerular filtration rate (eGFR) (mL/min/1.73m2) from baseline to Week 12 | At baseline, up to week 12
Absolute change in systolic blood pressure (SBP) (mmHg) from baseline to Week 12 | At baseline, up to week 12
Relative change (ratio) in Urine Albumin Creatinine Ratio (UACR) from baseline to Week 6 | At baseline, up to week 6
Absolute change in serum potassium (mmol/L) from baseline to Week 12 | At baseline, up to week 12

CONTACTS AND LOCATIONS:
Locations (159):
- United States (38):
  - Apogee Clinical Research, Huntsville, Alabama
  - Orange County Clinical Trials, Anaheim, California
  - North America Research Institute, San Dimas, California
  - Valiance Clinical Research-Tarzana-68237, Tarzana, California
  - Amicis Research Center - Valencia, Valencia, California
  - Focus Clinical Research, West Hills, California
  - Clinical Research of Brandon LLC, Brandon, Florida
  - Hillcrest Medical Research, DeLand, Florida
  - Encore Medical Research, Hollywood, Florida
  - Finlay Medical Research Corp, Miami, Florida
  - Total Research Group, LLC, Miami, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - West Orange Endocrinology, Ocoee, Florida
  - Florida Kidney Physicians - Riverview/Brandon, Riverview, Florida
  - Masters of Clinical Research, Inc, Augusta, Georgia
  - Velocity Clinical Research, Savannah, Savannah, Georgia
  - Boise Kidney and Hypertension, PLLC, Boise, Idaho
  - Research by Design, LLC, Chicago, Illinois
  - Nephrology Associates of Northern Illinois and Indiana - Oak Brook, Hinsdale, Illinois
  - Nephrology Associates of Northern Illinois and Indiana - Fort Wayne, Fort Wayne, Indiana
  - Kansas Nephrology Research Institute, LLC, Wichita, Kansas
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - Aa Mrc Llc, Flint, Michigan
  - Michigan Kidney Consultants, Pontiac, Michigan
  - Elixia MNA, LLC, City of Saint Peters, Missouri
  - Healor Primary Care, Las Vegas, Nevada
  - Endocrine Associates of Long Island, Smithtown, New York
  - Durham Nephrology Associates, Durham, North Carolina
  - Lucas Research, Inc., Morehead City, North Carolina
  - Brookview Hills Research Associates LLC, Winston-Salem, North Carolina
  - Heritage Valley Medical Group, Beaver, Pennsylvania
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Arlington Nephrology, Arlington, Texas
  - Endocrine Associates, Houston, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - Javara Inc.-Stephenville-68996, Stephenville, Texas
  - Utah Kidney Research Institute, Salt Lake City, Utah
  - Tidewater Physicians Multispecialty Group, Newport News, Virginia
- Argentina (6):
  - IDIM - Instituto de Diagnostico e Investigaciones Metabolicas, Buenos Aires
  - CEDIC - Centro de Investigacion Clinica, CABA
  - Mautalen- Salud e Investigacion, CABA
  - Sanatorio Güemes, Capital Federal
  - Instituto Medico Catamarca - IMEC, Rosario
  - CEMEDIC - Centro de Especialidades Medicas, Villa Luro
- Australia (4):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Austin Health, Heidelberg, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Belgium (4):
  - ULB Hopital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
  - Humani - CHU Charleroi - Chimay, Lodelinsart
- Brazil (8):
  - Centro de Pesquisa do Hospital Evangélico de Belo Horizonte, Belo Horizonte
  - Chronos Pesquisa Clinica, Brasília
  - Galileo Medical Research Ltda, Juiz de Fora
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
  - Cpquali Pesquisa Clinica Ltda, São Paulo
  - Fundação Oswaldo Ramos (Hospital do Rim), São Paulo
  - CEPIC - Centro Paulista de Investigacao Clinica, São Paulo
  - Centro de Pesquisa Clínica de Nefrologia do ICHC, São Paulo
- Canada (5):
  - Bluewater Clinical Research, Sarnia, Ontario
  - Heart Health Institute (Scarborough), Scarborough Village, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Diex Recherche (Trois-Rivieres), Trois-Rivières, Quebec
- China (15):
  - Beijing Tsinghua Changgung Hospital, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - NanFang Hosptial, Guangzhou
  - Zhejiang Province People's Hospital, Hangzhou
  - The Second Hospital of Anhui Medical University, Hefei
  - Center Hospital of Jinan, Jinan
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - The First People's Hospital of Nanning, Nanning
  - Ningbo Second Hospital, Ningbo
  - General Hospital of Ningxia Medical University, Ningxia
  - Second Hospital Affiliated to Shantou Medical University, Shantou
  - Shenzhen Second People's Hospital, Shenzhen
  - First Affiliated Hospital of Xi'an JiaoTong University, Xi'an
  - Yibin Second People's Hospital, Yibin
- Czechia (3):
  - DIKa centrum s.r.o., Havířov
  - MILAN KVAPIL s.r.o., Příbram
  - Nemocnice Slany, Slaný
- France (3):
  - HOP Bicêtre, Le Kremlin-Bicêtre
  - HOP Hôtel-Dieu, Nantes
  - HOP Civil, Strasbourg
- Germany (9):
  - Klinikum Bielefeld, Bielefeld
  - Internistische Gemeinschaftspraxis in Bünde, Bünde
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Frankfurt, Frankfurt
  - DaVita Clinical Research Germany GmbH Geilenkirchen, Geilenkirchen
  - Medizinische Hochschule Hannover, Hanover
  - Zentrum Für Nieren Hochdruck und Stoffwechselerkrankungen, Hanover
  - Nephrologische Gemeinschaftspraxis, Hamann/Bacinovic/Jacobsen, Rotenburg (Wümme)
  - Robert Bosch Gesellschaft für medizinische Forschung mbH, Stuttgart
- Italy (4):
  - Azienda Sanitaria Locale 2 Lanciano Vasto Chieti, Chieti
  - Università degli Studi di Perugia, Perugia
  - Istituto di Ricerche Farmacologiche Mario Negri IRCCS, Ranica (BG)
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
- Japan (8):
  - Kasugai Municipal Hospital, Aichi, Kasugai
  - National Hospital Organization Chibahigashi National Hospital, Chiba, Chiba
  - Tsuchiura Kyodo General Hospital, Ibaraki, Tsuchiura
  - Saiseikai Yokohamashi Nanbu Hospital, Kanagawa, Yokohama
  - Osaka General Medical Center, Osaka, Osaka
  - Ageo Central General Hospital, Saitama, Ageo
  - Omihachiman Community Medical Center, Shiga, Omihachiman
  - Tokyo Medical University Hachioji Medical Center, Tokyo, Hachioji
- Malaysia (3):
  - Hospital Canselor Tuanku Muhriz, Cheras
  - Tuanku Fauziah Hospital, Kangar
  - Hospital Kuala Lumpur, Kuala Lumpur
- Mexico (6):
  - Centenario Hospital Miguel Hidalgo, Aguascalientes
  - Unidad de Investigación Clinica y Atencion Medica HEPA SC, Guadalajara
  - Soltmed Smo, Mexico City
  - Clinica Omega Diabetes, Mexico City
  - Medical Care & Research SA de CV, Mérida
  - Sociedad de Metabolismo y Corazón S.C., Veracruz
- Netherlands (4):
  - Amsterdam UMC Locatie AMC, Amsterdam
  - Albert SchweitzerZiekenhuis, Dordrecht
  - Catharina Ziekenhuis, Eindhoven
  - Bethesda Diabetes Research Center, Hoogeveen, Hoogeveen
- New Zealand (3):
  - Momentum Clinical Research - Kapiti Coast, Kapiti, Wellington Region
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
- Philippines (4):
  - Norzel Medical and Diagnostic Clinic, Cebu City
  - Institute for Studies on Diabetes Foundation Inc., Marikina City
  - Philippine Heart Center, Quezon City
  - Senor Santo Nino Hospital, Tarlac City
- Poland (4):
  - Centrum Medyczne "Hipokrates" S.C. Elżbieta I Grzegorz Grześk, Bydgoszcz
  - American Heart Of Poland Sp. Z O.O., Chrzanów
  - Pro Familia Altera Sp. z o.o., Katowice
  - Pro Salus Sp. z o.o. sp.k., Lodz
- FDI Clinical Research - Mayagüez, Mayagüez, Puerto Rico
- South Korea (5):
  - Korea University Ansan Hospital, Ansan-si
  - Seoul National University Bundang Hospital, Seongnam
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wonju-si, Gangwon State
- Spain (6):
  - Centro de Salud Milladoiro, A Coruña
  - C.A.P. Sardenya, Barcelona
  - Centro de Salud Cartagena Casco Antiguo, Cartagena
  - Eap Osona Sud Alt Congost S.L.P. Cap Centelles, Centelles, Barcelona
  - Centro de Salud Naranco, Oviedo
  - Centro de Salud de San Juan, Salamanca
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
- Thailand (4):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakom Chiangmai Hospital, Chiang Mai
- United Kingdom (8):
  - University Hospital Monklands, Airdrie
  - Queen Elizabeth University Hospital, Glasgow
  - Belmont Health Centre, Harrow
  - Velocity Clinical Research, High Wycombe, High Wycombe
  - Richford Gate Medical Practice, London
  - Banbury Cross Health Centre, Oxford
  - Royal Berkshire Hospital, Reading
  - Sunderland Royal Hospital, Sunderland

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement'.For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor'spublication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency